CLINICAL TRIAL: NCT03510403
Title: Prospective Non-comparative Study to Assess the Efficacy, the Safety and the Acceptability of Nastent™ in Snoring and Obstructive Sleep Apnea Syndrome in European Population
Brief Title: Efficacy, Safety and Acceptability of Nastent™ in Snoring and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seven Dreamers Europe SAS (Industry)
Collaborators: Slb Pharma (Other); nastent.inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASTENT-17-FR
Record Dates: First submitted 2018-04-03; First posted 2018-04-27 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Snoring; Obstructive Sleep Apnea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device : nasal airway stent (Experimental): Patients with OSA or snoring use the nasal airway stent nastent™ each night for sleeping. The device is a tube-shaped medical device that is inserted from the nose and the tip of the tube reaches the soft palate. The inserted tube aids breathing by preventing the obstruction of the airway which causes poor sleep, frequent awakening during sleep and snoring.
  Interventions: Device: nastent™

INTERVENTIONS:
Device: nastent™ — Snorer and OSA patients (mild or moderate OSA) use the nasal airway stent for sleeping, each night for 1 month.

SUMMARY:
This study evaluates the efficacy, the tolerance and the acceptability/compliance of the nasal airway stent, Nastent, for the treatment of mild to moderate OSA and snoring in European adult patients without cardiovascular and/or respiratory comorbidities/disorders.

ELIGIBILITY:
Inclusion Criteria:

* Subject with newly diagnosed OSA (5≤AHI≤30 ev/h) or for whom treatment has failed (CPAP, mandibular repositioning device), or patients with snoring only (5<AHI)
* BMI≤30kg/m²
* Patient with good motivation to use the nasal device,
* Informed consent signed,
* Patient with social protection.

Exclusion Criteria:

* Cardiovascular comorbidities (resistant hypertension, recurrent atrial fibrillation, left ventricular failure, coronary heart disease and stroke),
* Respiratory comorbidities (respiratory failure, chronic obstructive pulmonary disease (COPD),
* Patient with one or more documented contraindication to use Nastent™,
* no regular partner,
* contraindication for sleep endoscopy,
* Psychiatric or neurological disorders (epilepsy),
* Progressive cancer or chronic inflammatory disease,
* AHI including more than 5 central apnea per hour,
* Allergy to one component of Nastent™.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Efficacy : change from baseline Snoring Intensity at 1 month | 1 month
  The snoring intensity will be evaluated by bed-partner of snorers and OSA patients using a Visual Analogue Scale (0-100 mm) at baseline and after 1 month of nastent™ use to assess the efficacy of treatment.
Efficacy : Change from baseline Apnea Hypopnea Index (AHI) at 1 month | 1 month
  The Apnea Hypopnea Index (number of apnea and hypopnea per hour) will be measured by respiratory polygraph on OSA patients subgroup at baseline and after 1 month of nastent™ use to assess the efficacy of treatment.

SECONDARY OUTCOMES:
Change from baseline Sleepiness at 1 month | 1 month
  The Epworth Sleepiness Scale (ESS) will be completed by OSA patients at baseline and after 1 month of nastent™ use to assess the evolution of somnolence/daytime sleepiness. Total score ranges between 0 and 24. A score above 10 indicates excessive daytime sleepiness.
Change from baseline Nasal Obstruction at 1 month | 1 month
  The NOSE questionnaire will be completed by snorers and OSA patients at baseline and after 1 month of nastent™ use to assess the efficacy of the device on the nasal obstruction.Total score ranges between 0 and 100.
Observance | 1 month
  The number of hours of Nastent™ use per night, the number of nights per week will be measured to assess the observance and compliance of the treatment in snorers and OSA patients during one month.
Adverse Events [Safety and Tolerability] | 1 month
  Adverse events reported by patient on a diary (from day 1 to day 30) and clinically observed by the physician will assess the safety and tolerability of the device.
Quality of Life using Functional Outcomes of Sleep Questionnaire (FOSQ-10) | 1 month
  FOSQ-10 measures functional status and difficulty in performing everyday activities via 10 questions. The questionnaire will be completed by snorer and OSA patients at baseline and after 1 month of nastent™ use to assess the evolution of the quality of life. Total score ranges between 5 and 20. Higher scores indicate better functional status.
Physician satisfaction | 1 month
  The physician's global satisfaction with nastent™ efficacy and safety will be assessed for each patient using a numeric scale after one month of treatment. Score ranges between 0 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Blumen, MD, Principal Investigator — Foch Hospital, Suresnes, FRANCE
Locations (6):
- France (6):
  - Cabinet ORL de Bordeaux, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Henri-Mondor Hospital, Créteil
  - Beau-Soleil Private Hospital, Montpellier
  - Centre Médical Veille Sommeil, Paris
  - Foch Hospital, Suresnes